CLINICAL TRIAL: NCT06443177
Title: The Effect of Sympathetic Modulation on Cerebral Vasospasm Secondary to Aneurysmal Subarachnoid Hemorrhage
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, Jesse G. A. Jones, MD, Assistant Professor, University of Alabama at Birmingham
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRB-300012920; UAB (Other: UAB)
Record Dates: First submitted 2024-05-06; First posted 2024-06-05 (Actual); Last update posted 2025-07-10 (Actual); Status verified 2025-07

CONDITIONS: Vasospasm, Cerebral; Aneurysmal Subarachnoid Hemorrhage
Keywords: aSAH; CVS; Sympathetic Modulation; Ruptured brain aneurysm
MeSH Terms: conditions — Vasospasm, Intracranial; Subarachnoid Hemorrhage

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Spinal Cord Stimulation (Experimental): Participants randomized to receive temporary electrode inserted through the skin into the epidural space of participants upper back/lower neck.
  Interventions: Device: Vectris trial leads and stimulation
- Sham Comparator (Sham Comparator): Participants randomized to not receive temporary electrode.
  Interventions: Device: Sham

INTERVENTIONS:
Device: Vectris trial leads and stimulation — The electrode is placed into the epidural space using standard epidural placement techniques with paramedian approach. The initial electrode settings have been adopted from prior studies. Should any significant discomfort be elicited from the stimulation, first the amplitude will be decreased to an acceptable level. If an acceptable level of stimulation is unable to be found, the stimulation will be discontinued.
  Arms: Spinal Cord Stimulation
Device: Sham — No electrode is placed.
  Arms: Sham Comparator

SUMMARY:
The purpose of the study is to see that in addition to existing therapy, how well an additional procedure named spinal cord stimulation might reduce blood vessel spasm from aneurysm rupture.

DETAILED DESCRIPTION:
The Investigators' overarching hypothesis is that sympathetic innervation plays a substantial role in conferring cerebral vasospasm (CVS) risk to aneurysmal subarachnoid hemorrhage (aSAH) patients and is associated with severity of clinical features and outcomes. Specifically, the Investigators surmise that central (hypothalamic) and local (arterial adventitia) sympathetic inputs are upregulated following SAH and integrate at the level of the neuromuscular junction to abnormally increase cerebrovascular tone. The long-term goal of this program is to use orthogonal approaches to undertake a comprehensive electrophysiological, functional genomics, and advanced imaging analysis of CVS. The Investigators hope is these data inform therapeutic pathways to modulate implicated pathogenic mechanisms and reduce CVS incidence and severity, thereby improving overall clinical outcomes in aSAH. In the short-term, the Investigators will focus on elucidating the modulatory role of cervical spinal cord stimulator (SCS) on sympathetic innervation to the cerebral vasculature.

This is a Phase 2 prospective, randomized single center study assessing the safety and efficacy of SCS for reducing vasospasm. aSAH patients who meet inclusion criteria and provide informed consent will be randomly assigned to SCS or a sham procedure. Subjects will be blinded until the end of the study, with no allowance for crossover. Temporary leads will stimulate, utilizing a paradigm established from prior human studies and the effect measured with daily transcranial doppler (TCD). Leveraging prior experience in vascular and functional neurosurgery, the Investigators' group is poised to make a substantial impact. Below the Investigators outline a feasible framework to modulate sympathetic drivers of CVS.

Aim 1: Perform feasibility analysis of SCS placement and operation in the aSAH setting. It is presently unknown how temporary SCS will impact the workflow and care of patients with acutely ruptured cerebral aneurysms. Given the rate of new aSAH cases at the Investigators' center (~50 per year), initiation of prospective data collection and longitudinal study are required. The Investigators will comprehensively assess operative time for electrode implantation, lead function and data transmission efficiency in the ICU, site infection/pressure injury and untoward systemic effects (hypotension, arrhythmia) for all patients enrolled at the Investigators' center.

Aim 2: Quantify the sympathetic modulating effect of SCS on cerebral blood flow during CVS. Further characterization of the sympathetic contribution to CVS will establish a rationale for functional/neuromodulatory therapies such as SCS. The Investigators will perform cervical epidural stimulation through temporary leads and monitor effects on cerebral blood flow by daily TCD. Experiments will continue throughout the 14-day CVS window to capture longitudinal changes in sympathetic tone and vascular response. Quantitative TCD metrics (velocity, resistance, Lindegaard ratio) will be compared between on- and off-stimulation epochs. The Investigators' study will not only fundamentally advance the Investigators' understanding of vasospasm, but also provide a framework to elucidate mechanisms of other cerebrovascular conditions.

ELIGIBILITY:
Inclusion Criteria:

1. Provision of signed and dated informed consent form
2. Stated willingness to comply with all study procedures and availability for the duration of the study
3. Diagnosed with Fisher grade 3 or 4 aneurysmal subarachnoid hemorrhage (1)
4. Ability to undergo endovascular treatment of aneurysmal subarachnoid hemorrhage
5. For females of reproductive potential: Negative pregnancy test at time of treatment
6. Plan to undergo standard of care and follow-up

Exclusion Criteria:

1. Medically unfit to undergo endovascular treatment (e.g., Hunt Hess grade 5)
2. Does not provide consent for the procedure.
3. Posterior circulation aneurysmal subarachnoid hemorrhage.
4. Initial aneurysm treatment after post bleed day 1

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2026-07-31 (Estimated); Primary Completion 2027-03-31 (Estimated); Study Completion 2027-07-31 (Estimated)

PRIMARY OUTCOMES:
Pre-Cerebrovascular response - Velocity | Day 1 - Day 14
  Pre-SCS measures of cerebral blood flow. Subjects will serve as their own internal control (on vs off stimulation) and be grouped collectively to enable more robust statistical analysis. To study the effect of SCS on cerebrovascular tone longitudinally over the course of the vasospasm window, mixed model statistics will be applied.
Pre-Cerebrovascular response - Resistance | Day 1 - Day 14
  Pre-SCS measures of cerebral blood flow. Subjects will serve as their own internal control (on vs off stimulation) and be grouped collectively to enable more robust statistical analysis. To study the effect of SCS on cerebrovascular tone longitudinally over the course of the vasospasm window, mixed model statistics will be applied.
Pre-Cerebrovascular response - Lindegaard ratio | Day 1 - Day 14
  Pre-SCS measures of cerebral blood flow. Subjects will serve as their own internal control (on vs off stimulation) and be grouped collectively to enable more robust statistical analysis. To study the effect of SCS on cerebrovascular tone longitudinally over the course of the vasospasm window, mixed model statistics will be applied.
Post-Cerebrovascular response - Velocity | Day 1 - Day 14
  Post SCS measures of cerebral blood flow. Subjects will serve as their own internal control (on vs off stimulation) and be grouped collectively to enable more robust statistical analysis. To study the effect of SCS on cerebrovascular tone longitudinally over the course of the vasospasm window, mixed model statistics will be applied.
Post-Cerebrovascular response - Resistance | Day 1 - Day 14
  Post SCS measures of cerebral blood flow. Subjects will serve as their own internal control (on vs off stimulation) and be grouped collectively to enable more robust statistical analysis. To study the effect of SCS on cerebrovascular tone longitudinally over the course of the vasospasm window, mixed model statistics will be applied.
Post-Cerebrovascular response - Lindegaard ratio | Day 1 - Day 14
  Post SCS measures of cerebral blood flow. Subjects will serve as their own internal control (on vs off stimulation) and be grouped collectively to enable more robust statistical analysis. To study the effect of SCS on cerebrovascular tone longitudinally over the course of the vasospasm window, mixed model statistics will be applied.
Transcranial Doppler (TCD) velocities of cerebral arteries | Day 1 - Day 14
  Daily transcranial Doppler studies will be performed to obtain quantitative data on cerebrovascular response during the critical 14-day vasospasm window.

SECONDARY OUTCOMES:
Overall Survival | Through study completion, approximately 24 months
  Overall survival is defined for all patients and measured from time of treatment to death or end of a study. The analyses for overall survival will be like that of the primary endpoint. It will also utilize Kaplan Meier methods and Cox proportional hazards modeling to compare the overall survival to the treatment-dependent prognosis index.

CONTACTS AND LOCATIONS:
Overall Officials: Jesse Jones, MD, Principal Investigator — University of Alabama at Birmingham
Locations (1):
- University of Alabama at Birmingham, Birmingham, Alabama, United States

IPD SHARING:
Plan to Share IPD: No